CLINICAL TRIAL: NCT00510939
Title: Phase II, Open-Label, Multi-centre, 2-part Study to Assess the Safety, Tolerability, and Efficacy of Tipifarnib Plus Bortezomib in the Treatment of Newly Diagnosed Acute Myeloid Leukemia (AML) Unfit for Conventional Chemotherapy ( >18 Years) or in Patients With Acute Myeloid Leukemia in First Relapse ( >60 Years)
Brief Title: Study to Assess the Safety, Tolerability, and Efficacy of Tipifarnib Plus Bortezomib in the Treatment of Acute Myeloid Leukemia
Acronym: HEMOS AML 0106
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Giovanni Martinelli, Dipartimento di Ematologia "Seragnoli"- Policlinico Sant'Orsola Bologna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEMOS AML 0106; EudraCT 2007-000273-35
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; NFkB activity and leukemia; expression of NFkB
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — tipifarnib; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tipifarnib plus Bortezomib

SUMMARY:
This is one of the first studies of combination of Zarnestra plus Velcade in man. A primary objective of the study is therefore to assess the safety and tolerability of multiple doses of Zarnestra plus Velcade in patients with AML.

New treatments for patients that are untreatable with intensive chemotherapy aged de novo AML patients or post-relapse AML are urgently required since, at present, many of the drugs used for second line therapy are the same as those used for first induction and response rates are much lower.

* The following evidence suggests that Velcade plus Zarnestra can be an attractive therapeutic combination for: AML patients.
* Affymetrix gene profiling data showed expression of NFkB1 in all of 5 myeloid cell lines cell lines tested and 35% of over 250 patient samples ( data generated in collaboration with Sergio Ferrari and Pier Paolo Piccaluga unpublished results, our Institute and University of Modena,Italy)
* Preclinical evidence showed that AML cells in suspension culture were prevented to develop de novo drug resistance and mediated drug resistance.

In Part B additional patients with AML will be treated to further characterize the tolerability,biological effects, and clinical efficacy of the combination Velcade plus Zarnestra. Patients on treatment for AML will undergo regular bone marrow aspirates and biopsies to assess responses to treatment. This will facilitate frequent assessment of biological endpoints (reduction in expression and phosphorylation of IKKb kinase, and downstream markers of signalling along with apoptosis, survival, proliferation and cellular size and ploidy) will be made in an attempt to confirm that the desired biological activity has been achieved at the maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Male or female aged >18 years with newly diagnosed Acute Myeloid Leukemia (AML), de novo or secondary, unfit for conventional chemotherapy
3. Male or female with Acute Myeloid Leukemia in first relapse ( > 60 years)
4. WHO performance status ³ 2, or/and unwillingness to receive conventional chemotherapy
5. Negative pregnancy test or evidence of post-menopausal status for female patients.
6. RASGRP1/APTX gene expression ratio calculated at the screening >10 (part B.2 only)

Exclusion Criteria:

1. Serum bilirubin 2 x> Upper Limit of Normal (ULN)
2. Aspartate aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT) >3.5 x ULN
3. Serum creatinine ³ 2.5 x ULN or 24-hour creatinine clearance £ 60 mL/min (measured or calculated by Cockcroft-Gault)
4. Patients with AML of FAB M3 classification (APL)
5. Patients with a history of another primary malignancy within the previous 1 year other than basal cell carcinoma or carcinoma in situ, the patient is in remission
6. Any clinically defined central nervous system AML.
7. Participation in an investigational drug study within the 30 days prior to entry
8. Evidence of uncontrolled infection or CNS-Hemorrhagic
9. Patients with documented cases of human immunodeficiency virus (HIV)
10. Peripheral Neuropathy or Neuropathic Pain grade > or = 2
11. Has known or suspected hypersensitivity or intolerance to boron, mannitol, or heparin, if an indwelling catheter is used
12. Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure (Attachment 7,NYHA Classification of Cardiac Disease), uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis
13. RASGRP1/APTX gene expression ratio calculated at the screening <10 (part B.2 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2007-03

PRIMARY OUTCOMES:
PART A: Assess the safety and tolerability of combined use of Zarnestra plus multiple ascending doses of Velcade in patients with de novo AML unfit for conventional chemotherapy (age >18 years) or in first or subsequent relapse ( >60 years).(COMPLETED) | August 2007
Part B.1: Assess the effect of Tipifarnib plus the defined in part A dose of Velcade in patients with de novo AML unfit for conventional chemotherapy (age >18 years) or in Patients in first or subsequent relapse ( >60 years) (COMPLETED) | December 2008
Part B.2: Evaluate the overall response (CR, PR, HI) of patients with a RASGRP1/APTX gene expression ratio > 10, identified as predictive of a good clinical response to tipifarnib in patients with de novo AML unfit for conventional chemotherapy. | June 2010

SECONDARY OUTCOMES:
To investigate the effect of Velcade on the expression of NFkB, and biomarkers of NFkB
Including phosphorylation of c-Rel on leukaemic blasts by flow cytometry, protein analysis,
Immunohistochemistry, and/or mRNA profiling using gene and SNPs DNA chip.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, MD, Principal Investigator — Istituto di Ematologia ed Oncologia Medica "L.eA.Seràgnoli" Policlinico S.Orsola-Malpighi di Bologna
Locations (1):
- Istituto di Ematologia "L e A Seragnoli" Policlinico S.Orsola-Malpighi, Bologna, Italy